CLINICAL TRIAL: NCT05740436
Title: POSTSCRIPTUM: Protocol of Geriatric Rehabilitation in Patients of 60 and Older Who Live in Moscow Boarding Houses or Nursing Homes. Protocol of Multicentral Prospective Study.
Brief Title: Protocol of Geriatric Rehabilitation in Patients of 60 and Older Who Live in Moscow Boarding Houses or Nursing Homes
Acronym: POSTSCRIPTUM
Status: Completed | Type: Observational
Sponsor: Pirogov Russian National Research Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/GR
Record Dates: First submitted 2023-02-13; First posted 2023-02-23 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Frail Elderly Syndrome
Keywords: geriatric rehabilitation; elderly; frailty; Complex geriatric assessment
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Frail elderly subjects: Frail subjects of 60 years and older will get geriatric rehabilitation program based on CGA
  Interventions: Other: Geriatric rehabilitation program based on CGA
- Pre-Frail elderly subjects: Pre-Frail subjects of 60 years and older will get geriatric rehabilitation program based on CGA
  Interventions: Other: Geriatric rehabilitation program based on CGA
- Non-frail elderly Frail subjects: Non-frail Frail subjects of 60 years and older will get geriatric rehabilitation program based on CGA
  Interventions: Other: Geriatric rehabilitation program based on CGA

INTERVENTIONS:
Other: Geriatric rehabilitation program based on CGA — Geriatric rehabilitation program based on CGA will be performed under physicians tight control for 21 days and will include physical activity, psychological training, diet correction, adaptation measures, polypragmasia correction.

SUMMARY:
After screening complex geriatric assessment (CGA) the participants will undergo geriatric rehabilitation programs. After termination of 21-day program, CGA will be repeated and subjects will get a program of long-term rehabilitation. A phone call in six months and a face-to-face visit in 12 months will be scheduled to follow-up and to evaluate the progress in rehabilitation.

DETAILED DESCRIPTION:
After screening complex geriatric assessment (CGA) the participants will undergo geriatric rehabilitation programs. The participation duration will not exceed 13.5 months including the screening period.

The study comprises three periods:

* screening (1-14 days)
* a treatment course of 21 days
* a follow-up period of 12 months On screening visit Study procedures will include
* Informed consent signing
* The Comprehensive Geriatric Assessment (CGA)
* The recommendations on a program of geriatric rehabilitation based on CGA

Visit 2 will be performed at the end of rehabilitation program. It will include:

* The abbreviated CGA
* The evaluation of the results of 21-days geriatric rehabilitation program
* The recommendations on a long-term geriatric rehabilitation

Visit 3 will be scheduled in 3 months after Visit 2 as a phone call. Special questionnaire will be suggested to study subjects. The questionnaire includes questions on implementation of a geriatric rehabilitation program and on quality of life

Visit 4- the last study visit will be performed in 12 months after Visit 2. It will include CGA and study completion procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 60 and older who wanted to participate in the study and signed a consent form.
2. One or more indications for geriatric rehabilitation:

   * A discharge after a hospitalization due to an acute illness (excluding stroke and myocardial infarction), trauma, surgery, including planned ones.
   * A condition leading to an acute impairment of functional status (stress, etc.)
   * Newly admitted patients
   * Abnormalities of gait and mobility (R26)

Exclusion Criteria:

1. One or more contraindications to geriatric rehabilitation:

   1. Severe sensory and cognitive impairment hampering rehabilitation
   2. End stage diseases requiring palliative care
   3. End stage frailty (bedridden patients)
2. An acute illness or an exacerbation of a chronic disease during two weeks before the enrollment in the study
3. A contradiction to any component of a rehabilitation program
4. Hearing or visual lost that can influence on study tests results
5. Refuse to participate in the study -

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 60 years old and older
Study Population: men and women aged 60 years and older eligible for geriatric rehabilitation, who were addmited to one of the study sites
Sampling Method: Non-Probability Sample
Enrollment: 420 (Actual)
Dates: Start 2021-08-21 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
functional status dynamics | 13 months
  Instrumental Activity Daily Life scale score

CONTACTS AND LOCATIONS:
Overall Officials: Olga N Tkacheva, Dr., Principal Investigator — - Pirogov Russian National Research Medical University, the Russian Research and Clinical Center for Gerontology
Locations (1):
- Russian Research and Clinical Center for Gerontology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No